CLINICAL TRIAL: NCT06239025
Title: Efficacy of Transversus Thoracis Muscle Plane Block in Patients Undergoing Cardiac Surgery. A Randomized Controlled Trial
Brief Title: Efficacy of Transversus Thoracis Muscle Plane Block in Patients Undergoing Cardiac Surgery
Acronym: TTMP_Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hôpital du Valais (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTMP
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: multimodal analgesia + ultrasound-guided Transversus Thoracis Muscle Plane Block with ropivacaine 0.5 % vs multimodal analgesia alone
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: syringes with the study drug will be prepared by a study nurse. the patient, investigators and all carers will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block + multimodal analgesia (Active Comparator): Multimodal analgesia + TTMP block with ropivacaine 0.5 %, 30 mL
  Interventions: Other: ultrasound-guided Transversus Thoracis Muscle Plane Block
- Multimodal Analgesia (No Intervention): Multimodal Analgesia without a block

INTERVENTIONS:
Other: ultrasound-guided Transversus Thoracis Muscle Plane Block — block with ropivacaine 0.5 %, 30 mL
  Arms: Block + multimodal analgesia

SUMMARY:
The goal of this randomized double blind study is to evaluate the analgesic efficacy of Transversus Thoracis Muscle Plane Block in patients undergoing cardiac surgery with median sternotomy.

one group of participants will receive multimodal analgesia plus ultrasound-guided Transversus Thoracis Muscle Plane Block with ropivacaine 0.5 % after induction of general anesthesia, the other group will receive multimodal analgesia without a bloc.

The investigators want to know if participants who receive the Transversus Thoracis Muscle Plane Block with ropivacaine have less pain than participants who do not receive a block.

DETAILED DESCRIPTION:
Participants who undergo elective cardiac surgery with median sternotomy are eligible. They will receive general anaesthesia with multimodal analgesia as is standard in our institution. For study purposes participants will be randomized in a double blinded fashion to receive a Transversus Thoracis Muscle Plane Block with 30 mL of ropivacaine 0.5 %, or no block. As the block is carried out after induction of general anesthesia the participants will not know to which group they are assigned.

all blocks will be carried out after induction of general anesthesia, under full sterile precautions, and with ultrasound guidance. multimodal analgesia intra- and postoperatively is standardized and consists of: sufentanil, ketamine, dexmedetomidine, dexamethasone, paracetamol, metamizole, IV morphine in ICU.

The investigators aim for fast track surgery, i.e. extubation either in the operating room or in ICU within the first 6 postoperative hours.

the primary outcome is postoperative opioid consumption over the first 24 h postoperatively, secondary outcomes are pain scores and opioid-related side effects. all outcomes will be assessed by blinded investigators.

ELIGIBILITY:
Inclusion Criteria:

* • Informed consent

  * Major adult (≥ 18 years old)
  * Body weight ≥ 50 kg. 50 kg is the minimal weight to ensure that participants will not receive an overdose of local anesthetic (ropivacaine 3 mg/kg)
  * Primary cardiac surgery via a sternotomy approach
  * Planned for fast-track procedure (i.e. postoperative extubation time of maximum six hours)

Exclusion Criteria:

* • Participation in another study within the 30 days preceding and during the present study

  * Refusal and/or inability to understand or sign the informed consent
  * Emergency cardiac surgery
  * Previous cardiac surgery
  * Hypersensitivity or allergy to ropivacaine and other amide-class LA
  * History of chronic pain
  * History of substance abuse
  * Severe cardiac dysfunction (i.e. LVEF ≤ 35%)
  * Severe obesity (BMI > 40kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
opioid consumption | 24 hours postoperatively
  cumulative intravenous morphine-equivalents

SECONDARY OUTCOMES:
Postoperative pain 2 h | 2 hours postoperatively
  Numeric Rating Scale 0-10
Postoperative pain 6 | 6 hours postoperatively
  Numeric Rating Scale 0-10
Postoperative pain 12 | 12 hours postoperatively
  Numeric Rating Scale 0-10
Postoperative pain 24 | 24 hours postoperatively
  Numeric Rating Scale 0-10
ICU length of stay | 5 days
  ICU length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital du Valais, Sion, Switzerland

IPD SHARING:
Plan to Share IPD: No